CLINICAL TRIAL: NCT01525888
Title: Renin-angiotensin-aldosterone System (RAAS) Blockade and Contrast Induced Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOR21711CTIL
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2012-01

CONDITIONS: Radiographic Contrast Agent Nephropathy
Keywords: Contrast induced nephropathy
MeSH Terms: interventions — Angiotensin Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): continue with treatment with angiotensin converting enzyme inhibitor or angiotensin blocker during all study period
- drug stop (Experimental): temporary stop of angiotensin converting enzyme inhibitor and angiotensin blocker treatment at least 72 hours before coronary angiography and renew of treatment 72 hours after angiography
  Interventions: Procedure: stop angiotensin converting enzyme inhibitor or angiotensin receptor blocker (ACE-I/ARB)

INTERVENTIONS:
Procedure: stop angiotensin converting enzyme inhibitor or angiotensin receptor blocker (ACE-I/ARB) — stoping for 6 days treatment with angiotensin converting enzyme inhibitor or angiotensin receptor blocker
  Arms: drug stop

SUMMARY:
The aim of the current study is to evaluate prospectively whether concomitant administration of renin-angiotensin-aldosterone system (RAAS) blockers (namely ACE-I and ARBs') influence the change in estimated glomerular filtration rate or GFR (eGFR) after administration of contrast media in patients undergoing non-emergent coronary angiography.

DETAILED DESCRIPTION:
Contrast-induced nephropathy (CIN) is defined as an absolute or relative increase in serum creatinine compared to the baseline values, together with exposure to a contrast agent and exclusion of alternative explanations for renal impairment. Most frequently the renal impairment develops 48 hours post exposure. Although RAAS blocking agents are widely used among patients requiring contrast studies, data regarding the effect of these agents on the development of CIN are sparse and inconsistent. Patients undergoing percutaneous coronary intervention are frequently treated with RAAS blocking agents. Despite the not infrequent occurrence of CIN following percutaneous coronary intervention (PCI) no guidelines are available on the topic of the cessation of the RAAS inhibitors prior to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years,
* chronic therapy with ACE-I and/or ARBs' (confirmed by electronic records in their medical file) and
* planned coronary angiography

Exclusion Criteria:

* chronic utilization of NSAIDS and Cox-2 selective inhibitors,
* chronic treatment with mineralocorticosteroid receptor blocker, and
* administration of contrast within 14 days prior to the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
change in eGFR from baseline to 48-72 hours following the exposure to the contrast. | 48 AND 72 HOURS AFTER EXPOSURE TO CONTRAST MEDIA